CLINICAL TRIAL: NCT04147338
Title: An Open-label, Randomized, Parallel-group Study to Assess the Pharmacokinetic Bioequivalence of Subcutaneously-administered Guselkumab Delivered by 3 Different Devices in Healthy Participants
Brief Title: A Study of Subcutaneously-administered Guselkumab Delivered by 3 Different Devices in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108698; CNTO1959CRD1003 (Other: Janssen Research & Development, LLC); 2020-003725-32 (EudraCT Number)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Reference Device: Guselkumab (Experimental): Participants will receive subcutaneous (SC) injections of guselkumab in reference device.
  Interventions: Drug: Guselkumab
- Test Device 1: Guselkumab (Experimental): Participants will receive SC injections of guselkumab in test device 1.
  Interventions: Drug: Guselkumab
- Test Device 2: Guselkumab (Experimental): Participants will receive SC injections of guselkumab in test device 2.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered subcutaneously.
  Other Names: CNTO 1959

SUMMARY:
The purpose of this study is to evaluate the serum concentration of guselkumab after administration using three different devices in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Have a weight in the range of 50.0 kilogram (kg) to 90.0 kg, inclusive
* Be healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening and Day -1. Any abnormalities must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* A female participant must have a negative pregnancy test result at screening and baseline (Day -1) and while enrolled in this study
* Contraceptive (birth control) use by men should be consistent with local regulations (if any) regarding the acceptable methods of contraception for those participating in clinical studies
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 12 weeks after study intervention

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal (GI) disease, neurologic or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* History of malignancy before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence
* Has a current chronic infection, prior history of recurrent infection, or an active infection
* Has previously received guselkumab
* Has a positive urine drug and alcohol screen during screening or at admission (Day -1)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Up to Day 85
  Cmax is the maximum observed serum concentration.
Area Under the Serum Concentration-Time Curve from Time Zero to Time Infinity (AUC [0-infinity]) | Up to Day 85
  AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinity time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the serum concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable concentration, and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 113 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are AEs which will occur up to 113 days that were absent before treatment or that worsened relative to pre-treatment state.
Number of Participants with Clinically Significant Vital Signs Abnormalities | Up to 113 days
  Number of participants with clinically significant abnormalities in the vital signs including temperature (oral), pulse rate, respiratory rate, and blood pressure will be reported.
Number of Participants with Clinically Significant Physical Examination Abnormalities | Up to 113 days
  Number of participants with clinically significant abnormalities in the physical examination (includes basic assessment of general appearance, respiratory and cardiovascular systems and the assessment of the skin at the administration area) will be reported.
Number of Participants with Clinically Significant Laboratory Abnormalities | Up to 113 days
  Number of participants with clinically significant abnormalities in laboratory assessments like serum chemistry, hematology, and urinalysis will be reported.
Number of Participants with Anti-Guselkumab Antibodies | Up to Day 85
  Number of participants with anti-drug antibodies to guselkumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Celerion, Tempe, Arizona, United States
- CRS Clinical Research Services, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency